CLINICAL TRIAL: NCT02433834
Title: A Randomized, Double-Blind, Chronic-Dosing (14 Days), 5-Period, 7-Treatment, Placebo-Controlled, Incomplete Block, Cross-Over, Multicenter, Dose-ranging Study to Assess the Efficacy and Safety of PT001 Relative to Placebo Metered Dose Inhaler and Open-Label Serevent® Diskus® in Adult Subjects With Intermittent Asthma or Mild to Moderate Persistent Asthma
Brief Title: Chronic Dosing Cross-Over Study to Assess the Efficacy and Safety of Glycopyrronium (PT001) in Adult Subjects With Intermittent Asthma or Mild to Moderate Persistent Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT001101-00
Record Dates: First submitted 2015-04-24; First posted 2015-05-05 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-05

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (7):
- GP MDI 28.8 μg (Experimental): GP MDI (PT001) 28.8 μg
  Interventions: Drug: Glycopyrronium MDI
- GP MDI 14.4 μg (Experimental): GP MDI (PT001) 14.4 μg
  Interventions: Drug: Glycopyrronium MDI
- GP MDI 7.2 μg (Experimental): GP MDI (PT001) 7.2 μg
  Interventions: Drug: Glycopyrronium MDI
- GP MDI 3.6 μg per (Experimental): GP MDI (PT001) 3.6 μg
  Interventions: Drug: Glycopyrronium MDI
- GP MDI 1.9 μg (Experimental): GP MDI (PT001) 1.9 μg
  Interventions: Drug: Glycopyrronium MDI
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Serevent® Diskus® 50 μg per inhalation (Active Comparator): Serevent® Diskus® 50 μg per inhalation
  Interventions: Drug: Serevent Diskus 50 μg

INTERVENTIONS:
Drug: Glycopyrronium MDI — GP MDI
  Arms: GP MDI 1.9 μg; GP MDI 14.4 μg; GP MDI 28.8 μg; GP MDI 3.6 μg per; GP MDI 7.2 μg
Drug: Serevent Diskus 50 μg
  Arms: Serevent® Diskus® 50 μg per inhalation
Drug: Placebo
  Arms: Placebo

SUMMARY:
A Randomized, Double-Blind, Chronic Dosing (14 days), 5-Period, 7-Treatment, Placebo-Controlled, Incomplete Block, Cross-Over, Multi-center, Dose-ranging Study to Assess the Efficacy and Safety of Glycopyrronium MDI (PT001) Relative to Placebo MDI and Open-Label Serevent Diskus in Adult Subjects With Intermittent Asthma or Mild to Moderate Persistent Asthma

ELIGIBILITY:
Inclusion Criteria:

1. Give their signed written informed consent to participate
2. Males and females ranging in age between 18 to 70 years, inclusive, before Screening (Visit 1a)
3. A female is eligible to enter and participate in the study if she is of: Non-child bearing potential (ie., physiologically incapable of becoming pregnant, including any female who is 2 years post-menopausal); or

   Child bearing potential, has a negative serum pregnancy test at Screening (Visit 1a), and agrees to 1 of the following acceptable contraceptive methods used consistently and correctly (ie., in accordance with the approved product label and the instructions of the physician for the duration of the study, from Screening [Visit 1a] until 14 days after Visit 12):
   * Complete abstinence from intercourse; or
   * Implants of levonorgestrel inserted for at least 1 month prior to the study drug administration, but not beyond the third successive year following insertion; or
   * Injectable progestogen administered for at least 1 month prior to study drug administration and administered for 1 month following study completion; or
   * Oral contraceptive (combined or progestogen only) administered for at least one monthly cycle prior to study drug administration; or
   * Double barrier method: condom or occlusive cap (diaphragm or cervical/vault caps) plus spermicidal agent (foam/gel/film/cream/suppository); or
   * An intrauterine device inserted by a qualified physician, with published data showing that the highest expected failure rate is less than 1% per year; or
   * Estrogenic vaginal ring; or
   * Percutaneous contraceptive patches
4. Asthma History: Have a diagnosis of intermittent asthma or mild to moderate persistent asthma, diagnosed at least 6 months prior to Screening (Visit 1a)
5. Reversibility: Diagnosis of asthma confirmed at Screening (Visits 1 and 2) with demonstration of reversibility to a bronchodilator defined as an FEV1 increase of at least 12% and at least 200 mL, 30 to 60 minutes after the inhalation of 4 puffs of salbutamol/albuterol (Ventolin HFA)
6. Pulmonary Function: Must have a pre-bronchodilator FEV1 ≥60% and ≤90% of predicted normal value at Visit 1a/b and Visit 2a/b
7. Asthma Maintenance Therapy: For those subjects receiving asthma maintenance therapy, they must be on a stable dose of ICS or non-ICS therapy (eg., LTRA) for at least 4 weeks prior to Screening (Visit 1a).
8. Results of clinical laboratory tests conducted at Screening (Visit 1a) must be acceptable to the Investigator.

Exclusion Criteria:

1. Life-Threatening Asthma: A subject must not have life-threatening asthma. Lifethreatening asthma is defined as a history of significant asthma episode(s) requiring intubation associated with hypercapnia, respiratory arrest, hypoxic seizures, or asthma related syncopal episode(s) within the 12 months prior to Visit 1a (Screening).
2. Worsening Asthma: A subject must not have experienced a worsening of asthma that involved an emergency department visit, hospitalization, or use of oral/parenteral corticosteroids within 6 weeks of Screening (Visit 1a).
3. Seasonal or Exercise-Induced Asthma Alone: Subjects with only seasonal or exerciseinduced asthma are excluded from participation.
4. Concurrent Respiratory Disease: A subject must not have current evidence or diagnosis of pneumonia, pneumothorax, atelectasis, pulmonary fibrotic disease, chronic bronchitis, emphysema, COPD, or other respiratory abnormalities other than asthma.
5. Concurrent Conditions/Diseases: A subject with historical or current evidence of any clinically significant, or comorbid or uncontrolled condition or disease state that, in the opinion of the Investigator, would put the safety of the subject at risk through study participation or would confound the interpretation of the results if the condition/disease exacerbated during the study.
6. Smoking History: Current smokers or former smokers who have stopped smoking within 6 months prior to enrollment or with a >10 pack year history of cigarettes, cigars, or pipe smoking. E-cigarettes and inhaled marijuana should be treated in the same manner as tobacco products.
7. Inhaled Anticholinergic Use: Subjects must not have used inhaled anticholinergics for at least the 2 weeks prior to Screening (Visit 1a).
8. Pregnant women or nursing mothers
9. Respiratory Tract Infection: Subjects who have had a respiratory tract infection within 6 weeks prior to Screening (Visit 1a). Subjects who develop a respiratory tract infection during the Screening Period must discontinue from the trial, but will be permitted to reenroll at a later date (at least 6 weeks after the resolution of the respiratory tract infection).
10. Uncontrolled Hypertension: Subjects who, in the opinion of the Investigator, have clinically significant uncontrolled hypertension.
11. Liver Function: Subjects with abnormal liver function tests defined as aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase, or total bilirubin ≥1.5 times the upper limit of normal on repeat testing.
12. Renal: a. Subjects with symptomatic prostatic hypertrophy that is clinically significant in the opinion of the Investigator (if treated and asymptomatic, the subject is eligible for enrollment). Subjects with a trans-urethral resection of prostate or full resection of the prostate within 6 months prior to Visit 1a are excluded from the study.

    b. Subjects with bladder neck obstruction or urinary retention that is clinically significant in the opinion of the Investigator. c. Subjects with a calculated creatinine clearance ≤30 mL/minute using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula [Levey, 2009] at Visit 1a and on repeat testing prior to Visit 3. Note: Subjects with overactive bladder syndrome treated with oral anticholinergics that have been on treatment for at least one month are allowed in the study.
13. Glaucoma: Subjects with a diagnosis of angle closure glaucoma will be excluded, regardless of whether or not they have been treated. Subjects with a diagnosis of glaucoma (non-angle closure), that in the opinion of the Investigator, has not been adequately treated will also be excluded. Subjects with previously diagnosed glaucoma who have intraocular pressure controlled with medication(s) are eligible. All medications approved for control of intraocular pressures are allowed including topical ophthalmic non-selective β-blockers such as betaxolol, carteolol, levobunolol, metipranolol, or timolol.
14. Cancer: Subjects who have cancer that has not been in complete remission for at least 5 years.

    Note: Subjects with squamous cell carcinoma and basal cell carcinoma of the skin that have been resected for cure are not considered exclusionary. Subjects with localized prostate cancer that in the opinion of the Investigator, has been adequately worked up, is clinically controlled, and the subject's participation in the study would not represent a safety concern, are eligible.
15. Drug Allergy: Subjects who have a history of hypersensitivity to lactose, milk proteins, or to any component of the MDI or dry powder inhaler (DPI)
16. Substance Abuse: Subjects with a known or suspected history of alcohol or drug abuse within the last 2-year period prior to Screening (Visit 1a).
17. Cardiac Conditions/Disease: Subjects with documented myocardial infarction within a year from the Screening (Visit 1a) are to be excluded. Subjects with a recent history of acute coronary syndrome, or who have undergone percutaneous coronary intervention or coronary artery bypass graft within 3 months of Screening (Visit 1a) are to be excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2015-05-27 (Actual); Primary Completion 2016-03-26 (Actual); Study Completion 2016-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shahid Siddiqui, Study Director — Pearl Therapeutics, Inc.
Locations (39):
- United States (39):
  - Pearl Therapeutics Inc., Birmingham, Alabama
  - Pearl Therapeutics Inc., Anaheim, California
  - Pearl Therapeutics Inc., Bakersfield, California
  - Pearl Therapeutics Inc., Cerritos, California
  - Pearl Therapeutics Inc., Los Angeles, California
  - Pearl Therapeutics Inc., Quartz Hill, California
  - Pearl Therapeutics Inc., Rancho Mirage, California
  - Pearl Therapeutics Inc., Rolling Hills Estates, California
  - Pearl Therapeutics Inc., Stockton, California
  - Pearl Therapeutics Inc., Colorado Springs, Colorado
  - Pearl Therapeutics Inc., Kissimmee, Florida
  - Pearl Therapeutics Inc., Miami, Florida
  - Pearl Therapeutics Inc., Ormond Beach, Florida
  - Pearl Therapeutics Inc., Evanston, Illinois
  - Pearl Therapeutics Inc., Iowa City, Iowa
  - Pearl Therapeutics Inc., Fall River, Massachusetts
  - Pearl Therapeutics Inc., North Dartmouth, Massachusetts
  - Pearl Therapeutics Inc., St Louis, Missouri
  - Pearl Therapeutics Inc., Omaha, Nebraska
  - Pearl Therapeutics Inc., Skillman, New Jersey
  - Pearl Therapeutics Inc., Verona, New Jersey
  - Pearl Therapeutics Inc., Asheville, North Carolina
  - Pearl Therapeutics Inc., Cornelius, North Carolina
  - Pearl Therapeutics Inc., Gastonia, North Carolina
  - Pearl Therapeutics Inc., Monroe, North Carolina
  - Pearl Therapeutics Inc., Raleigh, North Carolina
  - Pearl Therapeutics Inc., Shelby, North Carolina
  - Pearl Therapeutics Inc., Grove City, Ohio
  - Pearl Therapeutics Inc., Middleburg Heights, Ohio
  - Pearl Therapeutics Inc., Lake Oswego, Oregon
  - Pearl Therapeutics Inc., Medford, Oregon
  - Pearl Therapeutics Inc., Columbia, South Carolina
  - Pearl Therapeutics Inc., Dallas, Texas
  - Pearl Therapeutics Inc., El Paso, Texas
  - Pearl Therapeutics Inc., Killeen, Texas
  - Pearl Therapeutics Inc., McKinney, Texas
  - Pearl Therapeutics Inc., New Braunfels, Texas
  - Pearl Therapeutics Inc., San Antonio, Texas
  - Pearl Therapeutics Inc., Waco, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Randomized, Double-Blind, Chronic-Dosing (14 days), 5-Period, 7-Treatment, Placebo-Controlled, Incomplete Block, Cross-Over, Multi-Center, Dose-Ranging Study to Assess the Efficacy and Safety of PT001 Relative to Placebo MDI and Open-Label Serevent® Diskus® Adult Subjects With Intermittent Asthma or Mild to Moderate Persistent Asthma
Pre-assignment Details: Eligible subjects were randomized to 1 of 24 pre-defined treatment sequences. There were 5 treatment periods lasting 14 days with a 7-14 day washout period in between and a follow-up phone call 7-14 days post final dose. By-sequence tabulations of the data were not pre-specified.
Groups:
- Overall Study: All patients randomized
Period: Overall Study
Arm/Group | Overall Study
Started | 248
GP MDI 28.8 µg | 112
GP MDI 14.4 µg | 230
GP MDI 7.2 µg | 228
GP MDI 3.6 µg | 118
GP MDI 1.9 µg | 107
Placebo MDI | 174
SAL 50 µg | 167
Completed | 211 (Subject PT001101-040014 did not complete Period 4 but completed the study. CSR states 210 completed.)
Not Completed | 37
Not completed — Protocol-specified criteria | 7
Not completed — Protocol Violation | 3
Not completed — Lost to Follow-up | 6
Not completed — Withdrawal by Subject | 14
Not completed — Adverse Event | 6
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) Population is all patients randomized to treatment and used for Participant Flow. Modified ITT (MITT) population, a subset of ITT Population is all subjects treated, with post-treatment efficacy data from at least 2 treatment periods, no major protocol violation precluding the use of data, used for Baseline Characteristics
Arm/Group | Overall Study
Number analyzed (Participants) | 222
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.0 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142
  Male | 80

OUTCOME MEASURES:

1. Primary Outcome: Peak Change From Baseline in FEV1 Within 3 Hours Post-dosing on Day 15
Description: Forced Expiratory Volume in 1 second (FEV1) within 3 hours post-dosing on Day 15
Time Frame: From Day 1 to Within 3 hours post dosing on Day 15 in each of 5 treatment periods
Population: Modified Intent-to-Treat (mITT) population was a subset of the Intent-to-Treat (ITT) Population and included all subjects who received treatment, had post-treatment efficacy data from at least two treatment periods, and did not hav e a major protocol violation that would preclude the use of data from these periods.
Measure: Least Squares Mean (Standard Error); unit: Liter
Groups:
- GP MDI 28.8 µg: Glycopyrronium Metered Dose Inhaler (GP MDI) 28.8 µg
- GP MDI 14.4 µg: Glycopyrronium Metered Dose Inhaler (GP MDI) 14.4 µg
- GP MDI 7.2 µg: Glycopyrronium Metered Dose Inhaler (GP MDI) 7.2 µg
- GP MDI 3.6 µg: Glycopyrronium Metered Dose Inhaler (GP MDI) 3.6 µg
- GP MDI 1.9 µg: Glycopyrronium Metered Dose Inhaler (GP MDI) 1.9 µg
- Placebo MDI: Placebo MDI.
- SAL 50 µg: salmeterol 50 µg
Arm/Group | GP MDI 28.8 µg | GP MDI 14.4 µg | GP MDI 7.2 µg | GP MDI 3.6 µg | GP MDI 1.9 µg | Placebo MDI | SAL 50 µg
Number analyzed (Participants) | 101 | 212 | 202 | 109 | 99 | 158 | 155
Liter | 0.284 (0.0181) | 0.261 (0.0141) | 0.252 (0.0142) | 0.237 (0.0176) | 0.215 (0.0184) | 0.130 (0.0154) | 0.285 (0.0156)

2. Secondary Outcome: Change From Baseline in Morning Pre-dose Trough FEV1 on Day 15
Description: Change from baseline in morning pre-dose trough FEV1 on Day 15
Time Frame: Day 1-Day 15 in each of 5 treatment periods
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | GP MDI 28.8 µg | GP MDI 14.4 µg | GP MDI 7.2 µg | GP MDI 3.6 µg | GP MDI 1.9 µg | Placebo MDI | SAL 50 µg
Number analyzed (Participants) | 101 | 212 | 204 | 109 | 99 | 159 | 155
Liter | 0.073 (0.0165) | 0.047 (0.0116) | 0.042 (0.0118) | 0.012 (0.0159) | 0.018 (0.0168) | -0.012 (0.0133) | 0.059 (0.0135)

3. Secondary Outcome: FEV1 AUC0-3 on Day 15
Description: FEV1 AUC0-3 is the area under the curve for the change from baseline in FEV1 calculated using the trapezoidal rule. All observed data will be used with the trapezoidal rule to calculate AUC. To aid in interpretation, all AUC values will be normalized by dividing the AUC by the time from the first to the last non-missing value (typically 3 hours).
Time Frame: Day 1-Day 15 in each of 5 treatment periods
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liter
Arm/Group | GP MDI 28.8 µg | GP MDI 14.4 µg | GP MDI 7.2 µg | GP MDI 3.6 µg | GP MDI 1.9 µg | Placebo MDI | SAL 50 µg
Number analyzed (Participants) | 101 | 212 | 204 | 109 | 99 | 158 | 155
Liter | 0.191 (0.0170) | 0.167 (0.0131) | 0.146 (0.0133) | 0.147 (0.0165) | 0.113 (0.0173) | 0.038 (0.0144) | 0.190 (0.0146)

4. Secondary Outcome: Change From Baseline in Average Daily Pre-dose PEFR Over 14 Days
Description: Change from baseline in average daily pre-dose peak expiratory flow rate (PEFR) over 14 days Daily pre-dose PEFR and daily post-dose PEFR will each be calculated as the average of the AM and PM measurements recorded for a given day. If either the AM or PM assessment is missing, only the single measurement will be used. Analyses of average daily pre-dose PEFR, average daily post-dose PEFR, and rescue Ventolin HFA usage will use the average of the non-missing daily values recorded in the subject diaries over each week and over the last week of treatment within each period.
Time Frame: Day 1-Day 15 in each of 5 treatment periods
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | GP MDI 28.8 µg | GP MDI 14.4 µg | GP MDI 7.2 µg | GP MDI 3.6 µg | GP MDI 1.9 µg | Placebo MDI | SAL 50 µg
Number analyzed (Participants) | 105 | 209 | 205 | 108 | 97 | 158 | 152
L/min | 5.01 (4.947) | -6.54 (4.032) | -10.65 (4.052) | -2.98 (4.905) | -10.52 (5.130) | -22.57 (4.345) | -3.00 (4.417)

5. Secondary Outcome: Change From Baseline in Average Daily Post-dose PEFR Over 14 Days
Description: Daily pre-dose PEFR and daily post-dose PEFR will each be calculated as the average of the AM and PM measurements recorded for a given day. If either the AM or PM assessment is missing, only the single measurement will be used. Analyses of average daily pre-dose PEFR, average daily post-dose PEFR, and rescue Ventolin HFA usage will use the average of the non-missing daily values recorded in the subject diaries over each week and over the last week of treatment within each period.
Time Frame: Day 1-Day 15 in each of 5 treatment periods
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | GP MDI 28.8 µg | GP MDI 14.4 µg | GP MDI 7.2 µg | GP MDI 3.6 µg | GP MDI 1.9 µg | Placebo MDI | SAL 50 µg
Number analyzed (Participants) | 104 | 208 | 205 | 107 | 99 | 159 | 153
L/min | 5.53 (4.568) | -2.86 (3.790) | -5.38 (3.801) | 3.09 (4.530) | -5.68 (4.680) | -21.65 (4.041) | 3.55 (4.103)

6. Secondary Outcome: Change From Baseline in Average Daily Rescue Medication Use Over 14 Days
Description: as for outcome 5
Time Frame: Day 1-Day 15 in each of 5 treatment periods
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Puffs
Arm/Group | GP MDI 28.8 µg | GP MDI 14.4 µg | GP MDI 7.2 µg | GP MDI 3.6 µg | GP MDI 1.9 µg | Placebo MDI | SAL 50 µg
Number analyzed (Participants) | 107 | 210 | 209 | 109 | 100 | 161 | 154
Puffs | -0.42 (0.132) | -0.25 (0.105) | -0.24 (0.105) | -0.24 (0.131) | -0.23 (0.136) | -0.11 (0.114) | -0.63 (0.116)

7. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ-5) on Day 15
Description: The ACQ-5 measures 5 symptoms (woken at night by symptoms, wake in the morning with symptoms, limitation of daily activities, shortness of breath, and wheeze). The scale is 0-6, where 0=minimum and 6=maximum
Time Frame: Day 1-Day 15 in each of 5 treatment periods
Population: Modified Intent-to-Treat (mITT) population. The modified intent-to-treat (mITT) population included all randomized patients who received at least one dose of study drug. Patients were analyzed according to the treatment they received.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GP MDI 28.8 µg | GP MDI 14.4 µg | GP MDI 7.2 µg | GP MDI 3.6 µg | GP MDI 1.9 µg | Placebo MDI | SAL 50 µg
Number analyzed (Participants) | 106 | 215 | 211 | 110 | 101 | 160 | 158
Scores on a scale | -0.167 (0.0586) | -0.173 (0.0453) | -0.113 (0.0455) | -0.100 (0.0578) | -0.205 (0.0602) | -0.056 (0.0501) | -0.304 (0.0505)

ADVERSE EVENTS:
Time Frame: Adverse events captured from Day 1 through Final Follow up Visit, which is 7-14 days post last study drug dose, unless serious. If serious, they are captured from screening Visit 1 through Final Follow up Visit
Description: Safety Population includes all subjects who were randomized to treatment and received at least one dose of study treatment
Arm/Group | GP MDI 28.8 µg | GP MDI 14.4 µg | GP MDI 7.2 µg | GP MDI 3.6 µg | GP MDI 1.9 µg | Placebo MDI | SAL 50 µg
Serious Adverse Events (participants affected / at risk) | 0/112 | 0/230 | 0/228 | 0/118 | 0/107 | 1/174 | 0/167
Other Adverse Events (participants affected / at risk) | 9/112 | 15/230 | 16/228 | 8/118 | 8/107 | 13/174 | 9/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GP MDI 28.8 µg (N=112) | GP MDI 14.4 µg (N=230) | GP MDI 7.2 µg (N=228) | GP MDI 3.6 µg (N=118) | GP MDI 1.9 µg (N=107) | Placebo MDI (N=174) | SAL 50 µg (N=167)
Gastroenteritis, viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GP MDI 28.8 µg (N=112) | GP MDI 14.4 µg (N=230) | GP MDI 7.2 µg (N=228) | GP MDI 3.6 µg (N=118) | GP MDI 1.9 µg (N=107) | Placebo MDI (N=174) | SAL 50 µg (N=167)
Dry Mouth (Gastrointestinal disorders) | 9 (9) | 15 (15) | 16 (17) | 8 (8) | 8 (8) | 13 (13) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent it's opinions, or the opinions of the publication committee, if these differ with the proposed publication.